CLINICAL TRIAL: NCT00499681
Title: A Phase II Neo-Adjuvant Study of Letrozole in Combination With Lapatinib in Post -Menopausal Patients With HER2-Positive and Hormone Receptor-Positive Operable Breast Cancer
Brief Title: PhII Neo-Adjuvant Letrozole & Lapatinib in Pts w/HER2+ & Hormone Receptor+ Operable Breast CA SPORE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VICC BRE 0660; VU-VICC-BRE-0660; VU-VICC-061102; GSK-LAP107087
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive Lapatinib and Letrozole once daily for two weeks, following tumor measurement patients receive Lapatinib and Letrozole once daily for 14 weeks.
  Interventions: Drug: lapatinib ditosylate; Drug: letrozole
- Arm II (Experimental): Patients receive Letrozole and placebo once daily for 2 weeks, following tumor measurement patients receive Letrozole and Lapatinib once daily for 14 weeks.
  Interventions: Drug: lapatinib ditosylate; Drug: letrozole; Other: placebo

INTERVENTIONS:
Drug: lapatinib ditosylate — Given once daily, 1500mg, for 2 weeks; Given once daily, 1500mg, for 14 weeks in Arm II
  Other Names: GW572016
Drug: letrozole — Given once daily, 2.5mg, for 2 weeks; Given once daily, 2.5mg, for 14 weeks
  Other Names: Femara
Other: placebo — Given once daily for 2 weeks
  Arms: Arm II

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving letrozole together with lapatinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This randomized phase II trial is studying how well giving letrozole together with lapatinib works in treating postmenopausal women with stage I, stage II, or stage III breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the pathological complete response in patients with HER2-positive and hormone receptor-positive operable stage I-III breast cancer.

Secondary

* To determine tumor cell apoptosis in situ as measured by TUNEL analysis of tumor sections from fresh frozen or paraffin-embedded core biopsies. (Parts 1 and 2)
* To determine whether EGFR, P-EGFR, P-HER2, Ser118 P-ERα, P-Akt, and P-MAPK (by IHC using fresh frozen or paraffin-embedded core biopsies) predict the inhibition of proliferation in situ (Ki67) and/or induction of cell death (TUNEL). (Parts 1 and 2)
* To determine the safety profile of neoadjuvant letrozole and lapatinib. (Part 2)
* To evaluate tumor response to treatment as measured by ultrasound. (Part 2)
* To evaluate the rate of breast conservation surgery. (Part 2)
* To determine the inhibition in cell proliferation in situ in response to letrozole and lapatinib as measured by the change in percentage of Ki67-positive tumor cells (determined by IHC using tumor sections from fresh frozen or paraffin-embedded surgical material). (Part 2)

OUTLINE: This is a randomized, double-blind, placebo-controlled, two-part study.

* Part 1: Patients are randomized to treatment arm.

  * Patients receive lapatinib and letrozole once daily for 2 weeks.
  * Patients receive letrozole and placebo once daily for 2 weeks. Patients then proceed to part 2.
* Part 2: All patients receive lapatinib and letrozole once daily for 14 weeks. Patients then undergo surgical resection of disease.

Patients undergo tissue sample collection at baseline, at 2 weeks, and then at the time of surgery for biomarker and laboratory studies. Samples are analyzed by IHC and TUNEL.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion Criteria:

* Clinical stage I, II, or III operable invasive mammary carcinoma, confirmed by histological analysis

  * Measurable residual tumor at the primary site

    * Measurable disease is defined as any mass that can be reproducibly measured by physical examination, mammogram, and/or ultrasound and can be accurately measured in at least one dimension (longest diameter to be recorded) as 10 mm (1 cm)
* Available core biopsies from the time of diagnosis

  * May include sections of paraffin-embedded material
* Scheduled to undergo surgical treatment with either segmental resection or total mastectomy
* Prior history of contralateral breast cancer allowed if patient has no evidence of recurrence of their initial primary breast cancer within the last 5 years
* HER2-positive by Herceptest (3+) or FISH
* ER-positive and/or PR-positive by IHC

Exclusion Criteria:

* Locally recurrent breast cancer
* Evidence of distant metastatic disease (i.e., lung, liver, bone, or brain metastases)

PATIENT CHARACTERISTICS:

Inclusion Criteria:

* Female
* Postmenopausal, as defined by any of the following:

  * At least 55 years of age
  * Under 55 years of age and amenorrheic for at least 12 months OR follicle-stimulating hormone (FSH) values ≥ 40 IU/L and estradiol levels ≤ 20 IU/L
  * Prior bilateral oophorectomy or prior radiation castration with amenorrhea for at least 6 months
* ECOG performance status 0-1
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 1.5 times ULN
* Able to swallow and retain oral medication
* Cardiac ejection fraction normal by echocardiogram (or MUGA scan if an echocardiogram cannot be performed or is inconclusive)

Exclusion Criteria:

* Premenopausal breast cancer, pregnant, or lactating
* Serious medical illness, that in the judgment of the treating physician, places the patient at high risk of operative mortality
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel
* Ulcerative colitis
* History of other malignancy

  * Patients who have been disease-free for 5 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinomas are eligible
* Active or uncontrolled infection
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure

PRIOR CONCURRENT THERAPY:

Exclusion Criteria:

* Prior chemotherapy for primary breast cancer
* Tamoxifen or raloxifene as a preventive agent within the past 21 days
* Hormone replacement therapy (e.g., conjugated estrogens tablets [Premarin]) within the past month
* Prior therapy with anthracyclines
* Investigational drug within the past 30 days or 5 half-lives, whichever is longer
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, or any other biologic therapy) other than letrozole
* Concurrent treatment with an investigational agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open from 07/12/2007 through 12/09/2010.
Pre-assignment Details: This is a two-part study. Part I consists of two arms: investigational drug plus Letrozole or placebo and Letrozole. Part II is Letrozole plus Lapatinib. Six patients signed consent. Two patients had toxicity or relapse, thus withdrew from the study.
Groups:
- Lapatinib + Letrozole, Then Lapatinib + Letrozole: Part I: Some participants received Lapatinib 1500mg + Letrozole 2.5mg once daily (QD) for 2 weeks. Participants then underwent ultrasound imaging for tumor measurement, a core biopsy for molecular markers, and an optional FDG-PET/CT scan. Part II, participants received Lapatinib 1500mg + Letrozole 2.5mg QD for 14 weeks.
- Placebo + Letrozole, Then Lapatinib + Letrozole: Part I: some participants received Placebo + Letrozole 2.5mg once daily (QD) for 2 weeks. Participants then underwent ultrasound imaging for tumor measurement, a core biopsy for molecular markers, and an optional. FDG-PET/CT scan. Part II: participants received Lapatinib 1500mg + Letrozole 2.5mg QD for 14 weeks
Period: Overall Study
Arm/Group | Lapatinib + Letrozole, Then Lapatinib + Letrozole | Placebo + Letrozole, Then Lapatinib + Letrozole
Started | 4 | 2
Completed | 4 | 0
Not Completed | 0 | 2
Not completed — toxicity | 0 | 1
Not completed — disease progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib + Letrozole, Then Lapatinib + Letrozole | Placebo + Letrozole, Then Lapatinib + Letrozole | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 56.5 (1) | 74 (1) | 62 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pathological Complete Response
Description: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: at 14 weeks
Population: Participants who were available for measurement of response.
Measure: Number; unit: participants
Groups:
- Part I and Part II Letrozole Plus Laptinab: Participants received 2 weeks treatment with letrozole with lapatinib and 14 weeks treatment with letrozole and lapatinib
- Part 1: Letrozole Plus Placebo Part II Letrozole Plus Laptinab: Participants received 2 weeks treatment with letrozole with a placebo and 14 weeks treatment with letrozole and lapatinib
Arm/Group | Part I and Part II Letrozole Plus Laptinab | Part 1: Letrozole Plus Placebo Part II Letrozole Plus Laptinab
Number analyzed (Participants) | 4 | 2
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Lapatinib + Letrozole, Then Lapatinib + Letrozole | Placebo + Letrozole, Then Lapatinib + Letrozole
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib + Letrozole, Then Lapatinib + Letrozole (N=4) | Placebo + Letrozole, Then Lapatinib + Letrozole (N=2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib + Letrozole, Then Lapatinib + Letrozole (N=4) | Placebo + Letrozole, Then Lapatinib + Letrozole (N=2)
diarrhea (Gastrointestinal disorders) | 4 (8) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis, clinical exam (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis, functional/symptomatic (Gastrointestinal disorders) | 1 (1) | 0 (0)
dysgeusia (Renal and urinary disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 3 (7) | 1 (2)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
constitutional symptoms, other (General disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
rash, acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
skin/dermatology other (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
pain, other (General disorders) | 3 (3) | 0 (0)
pain, extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
pain breast (General disorders) | 1 (1) | 0 (0)
pain - NOS (General disorders) | 1 (1) | 0 (0)
pain, headache (General disorders) | 1 (1) | 0 (0)
hot flashes/flushes (Vascular disorders) | 1 (2) | 2 (2)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hemoglobn (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
leukocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
AST, SGOT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypoglycemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
depressed mood (Renal and urinary disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 2 (3) | 0 (0)
infection, bladder (Infections and infestations) | 1 (1) | 0 (0)
muscoloskeletal, soft tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
renal, burning (Renal and urinary disorders) | 0 (0) | 1 (1)
urinary, frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
gastrotestinal cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the restrictive nature of the eligibility criteria, only a total of 6 out of the planned 36 patients were accrued in 2 years, leading to early termination of the study. Hence, both clinical and correlative data were deemed uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes